CLINICAL TRIAL: NCT03542474
Title: Mild Cognitive Impairment and Endurance Exercise in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Rush University Medical Center (Other); Shirley Ryan AbilityLab (Other)
Responsible Party: Principal Investigator, Daniel Corcos, Professor of Physical Therapy and Human Movement Sciences, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU00202794
Record Dates: First submitted 2018-04-16; First posted 2018-05-31 (Actual); Results first posted 2020-07-14 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-06

CONDITIONS: Parkinson Disease; Mild Cognitive Impairment
MeSH Terms: conditions — Parkinson Disease; Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise (Experimental): 6 months of high intensity endurance exercise on a treadmill (3 times per week)
  Interventions: Behavioral: High Intensity Endurance Exercise

INTERVENTIONS:
Behavioral: High Intensity Endurance Exercise — Treadmill exercise at 80%-85% maximum heart rate for 30 minutes a day, 3 times per week, for 6 months.

SUMMARY:
The overall objective of this study is to determine how high intensity endurance exercise affects both cognition and the signs and symptoms of Parkinson's disease as well as if certain brain structures and functions also change with this exercise.

DETAILED DESCRIPTION:
The overall purpose and objective of this project is to test the hypothesis that high intensity endurance exercise causes beneficial brain adaptation in patients with mild cognitive impairment in Parkinson's disease (PD-MCI). Aim 1 will determine the effect of high intensity endurance exercise on cognitive function and other clinical symptoms in PD-MCI. Aim 2 will determine the effect of high intensity endurance exercise on brain structure and function in PD-MCI. Aim 3 will determine the effect of high intensity endurance exercise on cortisol in PD-MCI. Aim 4 will determine the effect of high intensity endurance exercise on inflammation-related biomarkers found in blood in PD-MCI. Aim 5 will determine the effect of high intensity endurance exercise on peripheral levels of neurotrophic factors found in blood in PD-MCI.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, ages 40-85
* A diagnosis of idiopathic PD
* A diagnosis of PD-MCI
* Due to the stringent head motion during fMRI, we will only include a patient with a head tremor of < 2.
* Hoehn and Yahr stage < or equal to 3
* Stable medication regimen for > or equal to 30 days before entering the study
* Living with a carepartner

Exclusion Criteria:

* PD subjects meeting MDS criteria for PD dementia or having a SCOPA-Cog score less than or equal to 16, or PD subjects having normal cognition defined as a SCOPA-Cog Score of is greater or equal to 25.
* Atypical or secondary parkinsonism as determined by referring Neurologist
* Other disorders that might interfere with ability to perform high intensity endurance exercise (e.g. history of stroke, respiratory problems, traumatic brain injury, known advanced osteoarthritis, or neuromuscular disease).
* Individuals with known injury, disease, or condition that would affect the ability to perform endurance exercise.
* Any other clinically significant medical condition, psychiatric condition, drug or alcohol abuse that would, in the judgment of the investigator, interfere with the subject's ability to participate in the study.
* "Vigorous athletes" participating in any exercise program 2X/week or more will be excluded.
* Individuals with any type of implanted electrical device (such as a cardiac pacemaker or a neurostimulator), or a certain type of metallic clip (i.e., an ° Persons who have had a long history of working in metal shops will be excluded unless they have had a previous orbital x-ray scan clearing them for participation in MRI studies.
* Females who are pregnant or might be pregnant will be excluded from participation.
* Individuals who are claustrophobic and unable to tolerate a brain MRI scan will be excluded.
* Treatment with cholinesterase inhibitors or memantine (i.e., medications approved for treatment of dementia) or medications affecting cognition (i.e., anticholinergics)
* Use of medications that might interfere with neuromuscular junction function such as D-penicillamine and aminoglycoside antibiotics.
* Use of medications that might interfere with the BOLD contrast or heart response to exercise (e.g. β blockers).
* Individuals at high risk for cardiovascular disease as defined in Table 2.2 by the new ACSM guidelines.(Medicine 2014)
* Younger than 40 and older than 85. We exclude participants younger than 40 because these young onset patients may not be typical of the majority of patients who get the disease later in life. We exclude participants older than 85 because of the limited evidence they can successfully complete a high-intensity endurance exercise program. We also exclude patients whose disease was diagnosed before the age of 40.
* Individuals with known endocrine abnormalities or steroid use that could affect cortisol levels (e.g., Cushing's syndrome, pituitary or adrenal gland disease or adrenalectomy, use of steroid-based medications.
* Individuals with strong history of chronic inflammatory or autoimmune diseases or history of chronic use of NSAIDs, which could cause abnormal levels of inflammatory markers in the plasma.
* We will exclude adults unable to consent, individuals who are not yet adults, pregnant women, prisoners and children from this study.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2018-11-05 (Actual); Study Completion 2019-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Corcos, PhD, Principal Investigator — Northwestern University; Jennifer Goldman, MD, Principal Investigator — Rush University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Exercise
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Exercise
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 7
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Cognitive Function
Description: Mean change in cognitive function from baseline to 6-months as measured by global statistical test (GST) for cognitive domains. This will be a composite score reported as Z-scores. The Z-score indicates the number of standard deviations away from the mean, which is based on normative (healthy control) data. A Z-score of 0 is equal to the mean of the normative data with negative numbers indicating values lower than the mean and positive values higher. A positive change in Z-scores indicates a favorable outcome.
  The GSTs will be calculated from the following neuropsychological tests administered in the cognitive test battery reflecting specific cognitive domains:
  * Attention/Working Memory - Trail Making Test-Part A
  * Executive Function - Trail Making Test-Part B, Clock Draw, Raven's Progressive Matrices
  * Memory - Hopkin Verbal Learning Test-Revised, Free and Cued Selective Reminding Test, Figural Memory Test
  * Processing Speed - Symbol Digit Modality Test
Time Frame: Baseline and 6 Months
Population: Raw scores for cognitive tests were transformed to Z-scores based upon normative data. Cognitive domain scores were calculated by averaging Z-scores for neuropsychological tests within specific domains, thereby accounting for any unequal distribution of tests per domain. Higher (more positive) scores indicate better outcome.
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Exercise
Number analyzed (Participants) | 8
z-score
  GST-Global Pre | -0.6960 (0.6691)
  GST-Global Post | -0.6095 (0.7506)
  GST-Attention/Working Memory Pre | 0.6018 (0.4147)
  GST-Attention/Working Memory Post | 0.6018 (0.4548)
  GST-Executive Function Pre | -1.657 (1.199)
  GST-Executive Function Post | -1.462 (1.240)
  GST-Memory Pre | -1.269 (0.7684)
  GST-Memory Post | -1.196 (0.7054)
  GST-Processing Speed Pre | -0.4596 (0.7840)
  GST-Processing Speed Post | -0.3820 (0.9025)

2. Secondary Outcome: 6 Month Change in Movement Disorder Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Total Score
Description: Mean change in total MDS-UPDRS score. This is a summed total from Part I (non-motor experiences of daily living), Part II (motor experiences of daily living, Part III (motor examination) and Part IV (motor complications). The minimum score on the MDS-UPDRS is 0 and the maximum is 260 with higher scores representing worse symptoms.
Time Frame: Baseline and 6 Months
Reporting Status: Not Posted

3. Secondary Outcome: 6 Month Change in Movement Disorder Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part II (Motor Experiences of Daily Living)
Description: Mean change in total MDS-UPDRS Part II (motor experiences of daily living) score. Part II comprises 13 items evaluating the impact of PD on patients' activities of daily living (ADL) over the week prior to the visit such as speech, salivation, swallowing, eating, handwriting, dressing, turning in bed, walking. The total score, being the sum of all these items, can be between 0 to 52. Higher scores represent worse symptoms.
Time Frame: Baseline and 6 Months
Reporting Status: Not Posted

4. Secondary Outcome: 6 Month Change in Movement Disorder Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part I Non Motor Experiences of Daily Living Score
Description: Mean change in total MDS-UPDRS Part I (non-motor experiences of daily living) score. Part I assesses 15 items of non-motor aspects of experiences of daily living. Part IA is assessed by a qualified rater, Part IB is completed by the patient. The total score, being the sum of all these items, can be between 0 to 60. Higher scores represent worse symptoms.
Time Frame: Baseline and 6 Months
Reporting Status: Not Posted

5. Secondary Outcome: 6 Month Change in Movement Disorder Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part IV Motor Complications Score
Description: Mean change in total MDS-UPDRS Part IV (motor complications) score. Part IV assesses motor complications of therapy, such as dyskinesias, motor fluctuations. This part (6 items) is completed by a qualified rater. The total score, being the sum of all these items, can be between 0 to 24. Higher scores represent worse symptoms.
Time Frame: Baseline and 6 Months
Reporting Status: Not Posted

6. Secondary Outcome: 6 Month Change in Movement Disorder Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Motor (Part III) Score
Description: Mean change in total MDS-UPDRS Part III (motor examination) score. The minimum score on the MDS-UPDRS Part III is 0 and the maximum is 132 with higher scores representing worse motor symptoms.
Time Frame: Baseline and 6 Months
Reporting Status: Not Posted

7. Secondary Outcome: 6 Month Change in Sleep Quality Evaluated by the Epworth Sleepiness Scale (ESS)
Description: The ESS assesses the overall level of daytime sleepiness. Eight items describe normative daily situations known to vary in their soporific qualities. Patients rate the likelihood of dozing off or falling asleep. The test is rated on a 4-point scale (0=would never doze off to 3=high chance of dozing off).
Time Frame: Baseline and 6 Months
Reporting Status: Not Posted

8. Secondary Outcome: 6 Month Change in Sleep Quality Evaluated by the Pittsburg Sleep Quality Index (PSQI)
Description: The Pittsburgh Sleep Quality Index (PSQI) contains 19 self-rated questions and 5 questions rated by the bed partner or roommate (if one is available). Only self-rated questions are included in the scoring. The 19 self-rated items are combined to form seven "component" scores, each of which has a range of 0-3 points.The global PSQI score is then calculated by totaling the seven component scores, providing an overall score ranging from 0 to 21, where lower scores denote a healthier sleep quality.
Time Frame: Baseline and 6 Months
Reporting Status: Not Posted

9. Secondary Outcome: 6 Month Change in Fatigue Evaluated by the Fatigue Severity Scale
Description: A 9-item questionnaire with questions related to how fatigue interferes with certain activities and rates its severity according to a self-report scale. The items are scored on a 7 point scale with 1 = strongly disagree and 7= strongly agree. The minimum score = 9 and maximum score possible = 63. Higher the score = greater fatigue severity.
Time Frame: Baseline and 6 Months
Reporting Status: Not Posted

10. Secondary Outcome: 6 Month Change in Mood Evaluated by the Hamilton Depression Scale (HAM-D)
Description: Although the HAM-D form lists 21 items, the scoring is based on the first 17. Eight items are scored on a 5-point scale, ranging from 0 = not present to 4 = severe. Nine are scored from 0-2. Higher scores represent more severe depression.
Time Frame: Baseline and 6 Months
Reporting Status: Not Posted

11. Secondary Outcome: 6 Month Change in Quality of Life Evaluated by the Parkinson Disease Neuro Quality of Life (Neuro-QOL)
Description: The NeuroQOL is a self-report of health related quality of life in 17 domains and sub-domains for adults. Item banks consist of 302 items in total (range from 5 to 45) which are used adaptively to test a variable number and content of items in a computer assisted testing format. All items are rated on a five option scale based on intensity (e.g. 1 = not at all, 2 = a little bit, 3 = somewhat, 4 = quite a bit, 5 = very much) or frequency ("never" to "always"). Raw scores are converted based on consistent metric (T-distribution) with data from the US general population with a T-score mean of 50 and standard deviation of 10.
Time Frame: Baseline and 6 Months
Reporting Status: Not Posted

12. Secondary Outcome: 6 Month Change in Quality of Life Evaluated by the Parkinson Disease Questionnaire 39 (PDQ-39)
Description: The PDQ-39 is a 39-item self-report questionnaire, which assesses Parkinson's disease-specific health related quality over the last month covering 8 dimensions 1) Mobility (10, #1-10) 2) Activities of daily living (ADL) (6, #11-16) 3) Emotional well-being (6, #17-22) 4) Stigma (4, #23-26) 5) Social support (3, #27-29) 6) Cognition (4, #30-33) 7) Communication (3, #34-36) 8) Bodily discomfort (3, #37-39) on a 5 point ordinal system (0=never, 4=always). Dimension score = sum of scores of each item in the dimension divided by the maximum possible score of all the items in the dimension, multiplied by 100. Each dimension total score range from 0 (never have difficulty) to 100 (always have difficulty). Lower scores reflect better QoL. Overall score can be summarized in the Parkinson's Disease Summary Index (PDSI) or PDQ-39 Summary Index (PDQ-39 SI).PDSI or PDQ-39 SI = sum of dimension total scores divided by 8.
Time Frame: Baseline and 6 Months
Reporting Status: Not Posted

13. Secondary Outcome: The Boston Naming Test
Description: The examiner begins with Item 1 and continues through Item 60, unless the patient is in distress or refuses to continue. The patient is told to tell the examiner the name of each picture and is given about 20 seconds to respond for each trial. The examiner writes down the patient's responses in detail, using codes. If the patient fails to give the correct response, the examiner at her or his discretion may give the patient a phonemic cue, which is the initial sound of the target word. After the patient completes the test, the examiner scores each item + or - according to the response coding and scoring procedures.
Time Frame: Baseline and 6 Months
Reporting Status: Not Posted

14. Secondary Outcome: Verbal Fluency Test
Description: The Verbal Fluency Test has two conditions, Letter Verbal Fluency and Category Verbal Fluency. Letter Verbal Fluency assesses the number of words beginning with certain letters that participants can generate within 60 seconds, the Category Verbal Fluency assesses the number of words within particular categories participants can generate within 60 seconds.
Time Frame: Baseline and 6 Months
Reporting Status: Not Posted

15. Secondary Outcome: Benton Judgement of Line Orientation Test
Description: Benton Judgment of Line Orientation Test is a standardized test with 30 items that is specific for visual spatial cognition. Tests will be administered at baseline, after 3, 6, 9 and 12 months of treatment.
  The minimum score is 0, indicating low visual spatial cognition. The maximum score is 30, indicating high visual spatial cognition
Time Frame: Baseline and 6 Months
Reporting Status: Not Posted

16. Secondary Outcome: Intersecting Pentagon Copying Test
Description: This involves the participant copying an intersecting double pentagon and is given a maximum score of 1 point based on the correctness of copying. The IPC addresses visuospatial constructional skills and executive function.
Time Frame: Baseline and 6 Months
Reporting Status: Not Posted

17. Secondary Outcome: Mini Balance Evaluation Systems Test
Description: Measure of dynamic balance, scores range from 0 (no Balance) to 28 good dynamic balance
Time Frame: Baseline and 6 Months
Reporting Status: Not Posted

18. Secondary Outcome: Timed Up and Go Test (TUG)
Description: This measures the time (in seconds) taken by a patient to rise to their feet from a sitting position, walk 3 metres in a straight line, turn around, walk back to the seat and sit down again
Time Frame: Baseline and 6 Months
Reporting Status: Not Posted

19. Secondary Outcome: Six Minute Walk Test
Description: Distance traveled during 6 minute walk
Time Frame: Baseline and 6 Months
Reporting Status: Not Posted

20. Secondary Outcome: Activities Specific Balance Confidence Scale
Description: The activities specific balance confidence scale is used to assess the level of fear of falling. It consists of 16 items reflecting the level of balance confidence from 0% (no confidence) to 100% (complete confidence)
Time Frame: Baseline and 6 Months
Reporting Status: Not Posted

21. Secondary Outcome: New Freezing of Gait Questionnaire
Description: The New Freezing of Gait Questionnaire (NFOG-Q) is a clinician-administered tool that aims to assess both the clinical aspects of FOG as well as its subsequent impairments on quality of life. The task ratings and scales are calculated into a summed NFOG-Q score. Part I detected the presence of FOG using a dichotomous item in which individuals were classified as a freezer (FR) or a non-freezer (NFR) if they had experienced FOG-episodes during the past month. Parts II and III were designed for FRs only, providing a total summed score between 0 and 28. Part II (items 2-6, scoring range 0-19) rated the severity of FOG based on its duration and frequency in its most common manifestation, i.e. during turning and initiation of gait. Part III rated the impact of FOG on daily life (items 7-9, scoring range 0-9). No separate on and off rating of parts II and III was considered to avoid unreliable assessment.
Time Frame: Baseline and 6 Months
Reporting Status: Not Posted

22. Secondary Outcome: 6 Month Change in Hippocampus Volumes on Structural MRI
Description: Change in hippocampus volumes on structural MRI
Time Frame: Baseline and 6 Months
Reporting Status: Not Posted

23. Secondary Outcome: 6 Month Change in Microstructural Integrity of White Matter Pathways on Diffusion Tensor Imaging
Description: Change in Microstructural integrity of white matter pathways on diffusion tensor imaging
Time Frame: Baseline and 6 Months
Reporting Status: Not Posted

24. Secondary Outcome: 6 Month Change in Functional Connectivity Among Brain Networks on Resting State fMRI
Description: Change in Functional connectivity among brain networks on resting state fMRI
Time Frame: Baseline and 6 Months
Reporting Status: Not Posted

25. Secondary Outcome: 6 Month Change in Salivary Cortisol Levels
Description: Change in salivary cortisol levels between baseline and 6 months post exercise. Cortisol samples were taken before the exercise intervention (Pre) and after the exercise intervention (Post) at 8 different time points: At awakening (0), 15 minutes post awakening (0.25), 30 minutes post awakening (0.5), 45 minutes post awakening (0.75), 3 hours post awakening (3), 6 hours post awakening (6), 9 hours post awakening (9), and 12 hours post awakening (12).
Time Frame: Baseline and 6 Months
Measure: Mean (Standard Error); unit: nmol/l
Arm/Group | Exercise
Number analyzed (Participants) | 8
nmol/l
  0 Pre | 13.064 (2.1)
  0 Post | 10.486 (1)
  0.25 Pre | 18.996 (2.6)
  0.25 Post | 15.568 (1.5)
  0.5 Pre | 18.196 (2.2)
  0.5 Post | 16.29 (1.9)
  0.75 Pre | 19.34 (2.6)
  0.75 Post | 14.247 (1.4)
  3 Pre | 12.693 (3)
  3 Post | 6.711 (0.8)
  6 Pre | 5.301 (0.66)
  6 Post | 5.48 (0.7)
  9 Pre | 4.831 (0.7)
  9 Post | 4.525 (0.3)
  12 Pre | 3.233 (0.57)
  12 Post | 3.083 (0.4)

26. Secondary Outcome: 6 Month Change in Soluble Inflammatory Biomarkers in Plasma
Description: Change in soluble inflammatory biomarkers in plasma between baseline and 6 months post exercise
Time Frame: Baseline and 6 Months
Reporting Status: Not Posted

27. Secondary Outcome: 6 Month Change in Peripheral Levels of Neurotrophic Factors in Plasma
Description: Change in peripheral levels of neurotrophic factors in plasma between baseline and 6 months post exercise
Time Frame: Baseline and 6 Months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Exercise
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 4/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Exercise (N=8)
Fall (Injury, poisoning and procedural complications) | 2
Back pain (Injury, poisoning and procedural complications) | 1
Outpatient surgery (Surgical and medical procedures) | 1
Hip Pain (Injury, poisoning and procedural complications) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-06): https://cdn.clinicaltrials.gov/large-docs/74/NCT03542474/Prot_SAP_000.pdf